CLINICAL TRIAL: NCT07318285
Title: A Modified Technique of Target Lidocaine Infusion for Pain Control in Office Hysteroscopy: A Double-Blind Randomized Controlled
Brief Title: Targeted Lidocaine Infusion for Pain Reduction in Office Hysteroscopy
Acronym: OPTILID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: YAARA TABIB (Other)
Responsible Party: Sponsor-Investigator, YAARA TABIB, Principal Investigator, Obstetrics and Gynecology Research Unit, Hadassah Medical Center, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0220-25-HMO
Record Dates: First submitted 2025-11-30; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Hysteroscopy / Methods; Lidocaine Infusion; Placebo - Control
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Participants in this arm will receive 5 mL of normal saline infused through the internal cervical os immediately before office hysteroscopy.
  Interventions: Other: Saline (0.9% NaCl)
- Lidocaine Group (Experimental): Participants in this arm will receive 5 mL of 2% lidocaine infused through the internal cervical os immediately before office hysteroscopy.
  Interventions: Drug: Lidocaine %2 ampoule

INTERVENTIONS:
Drug: Lidocaine %2 ampoule — A 5 mL dose of 2% lidocaine solution will be infused slowly through the internal os using the hysteroscope before the start of uterine cavity distension.
  Arms: Lidocaine Group
Other: Saline (0.9% NaCl) — A 5 mL dose of sterile normal saline will be infused slowly through the internal os using the same technique as in the intervention arm, immediately before cavity distension.
  Arms: Control Group

SUMMARY:
The goal of this study is to find out whether a small amount of lidocaine (a common local anesthetic) can reduce pain during office hysteroscopy - a procedure used to look inside the uterus. The study will compare lidocaine to saline (salt water) to see which one helps more with pain relief.

Participants will:

1. Receive either lidocaine or saline gently applied inside the cervix right before the procedure
2. Undergo the hysteroscopy as planned
3. Be asked to rate their pain and satisfaction after the procedure

Lidocaine is commonly and safely used in dental and gynecological procedures. Participation is voluntary, and the procedure itself will not change.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Referred for outpatient diagnostic or operative (see-and-treat) hysteroscopy
* Able and willing to provide written informed consent

Exclusion Criteria:

* Pregnancy
* Active pelvic inflammatory disease or cervicitis
* Inability to consent
* Anti-psychotic drugs usage
* Previews cervical surgery (i.e., conization).
* Any contraindication for office hysteroscopy- cervical malignancy, profuse uterine bleeding, invisible external os, recent uterine perforation.
* Known allergy or hypersensitivity to Lidocaine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain During Hysteroscopy Procedure Assessed by Visual Analog Scale (VAS) | Immediately during the hysteroscopy procedure
  Pain experienced during the procedure, evaluated using a Visual Analog Scale (VAS). The VAS score ranging between 0 (no pain) to 10 (worst imaginable pain). Subgroup analyses will be performed by age group, parity, cesarean delivery history, and menopausal status.
Number of Participants with Successful Access to the Uterine Cavity | During the hysteroscopy procedure
  The number of participants for whom hysteroscopy successfully reached the uterine cavity, without the need to stop or repeat the procedure.
  This binary outcome (Yes/No) will be assessed by the performing physician during the procedure. Subgroup analyses will be performed by age group, parity, cesarean delivery history, and menopausal status.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Pain Score 5 Minutes After the Procedure | 5 minutes after completion of the hysteroscopy procedure
  Pain intensity assessed using a Visual Analog Scale (VAS) exactly 5 minutes following the end of the hysteroscopy. The VAS score ranging between 0 (no pain) to 10 (worst imaginable pain). Subgroup analyses will be performed by age group, parity, cesarean delivery history, and menopausal status.
Change in Visual Analog Scale (VAS) Pain Score from Baseline to During the Procedure | Changes of VAS score of pain from baseline (before procedure) and at 5 minutes of during procedure.
  The outcome will measure the change in pain score using the Visual Analog Scale (VAS) from baseline (immediately before the hysteroscopy) to during the procedure. The VAS score ranging between 0 (no pain) to 10 (worst imaginable pain). Subgroup analyses will be performed by age group, parity, cesarean delivery history, and menopausal status.
Completed procedure | During the hysteroscopy procedure
  Successful performance of the intended hysteroscopic procedure. Subgroup analyses will be performed by age group, parity, cesarean delivery history, and menopausal status.
Patient satisfaction | Immediately after the procedure
  Patient-reported satisfaction with the procedure using a validated 5-point Likert scale. Subgroup analyses will be performed by age group, parity, cesarean delivery history, and menopausal status.
Adverse effect | During and up to 10 minutes after the procedure
  Recording any vasovagal symptoms observed or reported, including nausea, bradycardia, or hypotension.

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results of the primary and secondary outcomes reported in any publication will be shared in anonymized format. Data will include coded patient level information and the data dictionary. Identifiable information will not be shared. Data will be available to qualified researchers upon request following publication of study results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available starting 6 months after publication and for a period of 5 years
Access Criteria: Access will be granted to researchers with approved scientific proposals. Requests will be reviewed by the principal investigator and institutional review board. Data will be shared through secure institutional channels.

REFERENCES:
- [Background] Barel O, Preuss E, Stolovitch N, Weinberg S, Barzilay E, Pansky M. Addition of Lidocaine to the Distension Medium in Hysteroscopy Decreases Pain during the Procedure-A Randomized Double-blind, Placebo-controlled Trial. J Minim Invasive Gynecol. 2021 Apr;28(4):865-871. doi: 10.1016/j.jmig.2020.08.003. Epub 2020 Aug 14. PMID 32798723
- [Background] Shankar M, Davidson A, Taub N, Habiba M. Randomised comparison of distension media for outpatient hysteroscopy. BJOG. 2004 Jan;111(1):57-62. doi: 10.1046/j.1471-0528.2003.00004.x. PMID 14687053
- [Background] Sagiv R, Sadan O, Boaz M, Dishi M, Schechter E, Golan A. A new approach to office hysteroscopy compared with traditional hysteroscopy: a randomized controlled trial. Obstet Gynecol. 2006 Aug;108(2):387-92. doi: 10.1097/01.AOG.0000227750.93984.06. PMID 16880310